CLINICAL TRIAL: NCT06582576
Title: Investigation of the Putative Mechanisms Underlying the Symptom-lowering Effect of the Enterra Medical Gastric Electrical Stimulator for Gastroparesis Treatment
Brief Title: Mechanisms of Action for the Enterra Medical Gastric Electrical Stimulator
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aalborg University Hospital (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GES - mechanisms of action
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Gastroparesis; Vomiting; Nausea
MeSH Terms: conditions — Gastroparesis; Vomiting; Nausea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Responders: Individuals who have a gastric pacemaker for treating gastroparesis and have experienced a "substantial or full" symptomatic improvement after the implantation.
  Interventions: Diagnostic Test: Effect of different gastric electrical stimulator stimulation paragdimes on brain, heart, and stomach.
- Non-responders: Individuals who have a gastric pacemaker for treating gastroparesis and answered have experienced "some or none" symptomatic improvement after the implantation.
  Interventions: Diagnostic Test: Effect of different gastric electrical stimulator stimulation paragdimes on brain, heart, and stomach.

INTERVENTIONS:
Diagnostic Test: Effect of different gastric electrical stimulator stimulation paragdimes on brain, heart, and stomach. — Measuring EEG, ECG, and ultrasound in both groups during different stimulation intensities provided by the previously implanted gastric electrical stimulator.

SUMMARY:
Background: Gastric electrical stimulation applied by a surgically implanted device effectively alleviates upper gastrointestinal symptoms in the majority of individuals with medically refractory gastroparesis. Despite its efficacy, the mechanisms of action have been minimally explored in previous studies, and it is unknown why some individuals experience limited symptom-lowering effects.

Aim: The investigators aim to investigate two of the potential mechanisms of action leading to symptom-reducing effects of gastric electrical stimulation: 1) possible central effects in the brainstem and brain by enhanced parasympathetic vagal activity, and 2) peripheral effects in the stomach by improved gastric accommodation.

Methods: Up to thirty individuals with drug-refractory gastroparesis having an implanted gastric electrical stimulator will be enrolled in this cross-sectional and observational study. Of these, 15 will be responders (substantial symptomatic improvement) and 15 non-responders (minor symptomatic improvement). Electroencephalography (EEG) will evaluate the stimulation-induced activity in the brain and brainstem to assess whether the gastric stimulation generates evoked potentials. Electrocardiography (ECG) will investigate stimulation-induced changes in the autonomic regulation of the heart. Gastric ultrasound will investigate the effect of stimulation on stomach accommodation, contractions, and wall tension. These central and peripheral measures will be assessed during one study day before and after activating the gastric electrical stimulator, following an increase in stimulation intensity and post-meal consumption. Furthermore, results will be compared between responders and non-responders.

Perspectives: Adjusting the parameters of gastric electrical stimulation based on objective markers in the brain, heart, or stomach, rather than relying on symptom fluctuations, may enhance the effectiveness of symptom improvement. In the future, these objective markers may aid in differentiating between responders and non-responders, which may lead to optimised selection criteria for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Able to read and understand Danish
* Have an implanted gastric electrical stimulator for treating gastroparesis
* Answering 0 or 1 (non-responders) or 3 or 4 (responders) on the Likert scale describing the symptom improvement gained by gastric electrical stimulation.
* Personally signed and dated the informed consent documents ("Informeret samtykke") indicating that the patient has been informed of all pertinent aspects of the trial
* Are willing and able to comply with the scheduled visit and trial procedures

Exclusion Criteria:

* Previous surgery on the vagus nerve, including cervical vagotomy
* Prior thoracic, abdominal or brain surgeries that, in the opinion of the investigator, could limit data collection or interpretation.
* Previous diagnosis or history of orthostatic intolerance, e.g. POTS, neurocardiogenic syncope, orthostatic hypotension or autonomic dysfunction.
* Patients with an implanted cardiac device (e.g. pacemaker, CRT, etc.) or vagal nerve stimulator (VNS).
* History of neurological disease that, in the opinion of the investigator, could limit data collection or interpretation.
* Participants with any clinical abnormalities that, in the opinion of the investigator, may increase the risk associated with trial participation or may interfere with the interpretation of the trial results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals having an implanted Enterra gastric electrical stimulator for treating gastroparesis. 15 will be included as "responders" and 15 as "non-responders". Using a 5-point Likert scale, each participant will evaluate the experienced symptom-reducing effect of the gastric electrical stimulation. The individuals answering 0 or 1 (minor or no symptom improvement) are defined as responders, while individuals answering 3 or 4 (substantial or full symptom improvement) are defined as responders. Individuals answering 2 will not be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Evoked brain potentials | 5min during maximum stimulation intensity
  Amplitude of evoked brain potentials induced by gastric electrical stimulation

SECONDARY OUTCOMES:
EEG measures between ON/OFF stimulation | 5min
  EEG frequency distribution when comparing the OFF and ON stimulation modes
Meal-related EEG measures | 5min
  EEG frequency distribution in response to an ingested meal when comparing the OFF and ON stimulation modes.
ECG measures between ON/OFF stimulation | 5min
  Heart rate variability, periodic repolarisation dynamic, and the deceleration capacity of the heart rate when comparing the OFF and ON stimulation modes.
ECG measures between stimulation intensities | 5min
  Heart rate variability, periodic repolarisation dynamic, and the deceleration capacity of the heart rate following different stimulation intensities.
Meal-related ECG measures | 5min
  Heart rate variability, periodic repolarisation dynamic, and the deceleration capacity of the heart rate in response to an ingested meal when comparing the OFF and ON stimulation modes.
Meal-related gastric accomodation | 5min
  Gastric accommodation in response to an ingested meal comparing OFF and ON stimulation.
Meal-related gastric tension | 5min
  Gastric tension in response to an ingested meal comparing OFF and ON stimulation.
Meal-related gastric contraction frequency | 5min
  Gastric contraction frequency in response to an ingested meal comparing OFF and ON stimulation.
Symptoms and gastric measures | 5min
  Correlation between gastroparesis symptoms (Gastroparesis Cardinal Symptom Index) and changes in gastric accommodation/tension when turning the stimulation ON after meal ingestion.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of hepatology and gastroenterology, Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No
The final dataset can be provided upon reasonable request